CLINICAL TRIAL: NCT00321659
Title: Short and Long-term Effects of Exercise and Education as Self-management in Women With Fibromyalgia
Brief Title: Optimizing Fibromyalgia Self-management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Arthritis Foundation (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Daniel Rooks, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001P001769; K23AR048305 (NIH)
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; self-management; exercise; patient education
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic and flexibility exercise (Experimental): 16 weeks of aerobic and flexibility exercise. Three days per week for 1 hour of walking and cycling.
  Interventions: Behavioral: Aerobic
- Strength, aerobic, and flexibility (Experimental): 16 weeks of strength training, aerobic, and flexibility exercise (ST) intervention;
  Interventions: Behavioral: Strength training
- Fibromyalgia Self-Help Course (Experimental): 7 weeks of FSHC behavior change education
  Interventions: Behavioral: FSHC
- a Combination of ST and FSHC (Experimental): 16 wks of a combination of ST and FSHC (ST-FSHC) exercise and behavior change education
  Interventions: Behavioral: Combination

INTERVENTIONS:
Behavioral: Aerobic — 3x/week of walking and cycling
  Arms: Aerobic and flexibility exercise
Behavioral: Strength training — 3x/week of resistance training activities
  Arms: Strength, aerobic, and flexibility
Behavioral: Combination — 3x/week of aerobic and strength training activities
  Arms: a Combination of ST and FSHC
Behavioral: FSHC — Biweekly group education group meetings
  Other Names: Fibromyalgia Self-Help Course
  Arms: Fibromyalgia Self-Help Course

SUMMARY:
The overall objective of this work is to improve treatment outcomes for persons with fibromyalgia by optimizing the approach to self-management. The purpose of this research project is to evaluate and compare, in a randomized, controlled trial involving 200 women, the short and long-term effectiveness of four approaches to fibromyalgia self-management for improving health and functional status, self-efficacy, and symptom severity. Additionally, we will also examine the effect of each intervention on health care usage. We will assess the following 16-week interventions:

* cardiovascular and flexibility exercise
* strength training, cardiovascular and flexibility exercise
* Arthritis Foundation's Fibromyalgia Self-Help course
* a combination of the Fibromyalgia Self-Help Course and strength training exercise interventions

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a common, chronic musculoskeletal disorder and a growing cause of disability and increased health care utilization. Current treatment focuses largely on pharmacological interventions, which are often ineffective at improving symptoms and functional status. Recent research suggests that disease self-management can be efficacious in the short-term at reducing symptom severity and improving function in persons with FMS. The most common forms of FMS self-management are coping skills training (behavioral/education) and exercise. Limited in number, most FMS self-management studies examine the short-term effects of one form or the other, with most using the coping skills training approach. Little data exist to examine the long-term effects of these interventions, the potential additive effect of combining coping skills training with a comprehensive, group exercise program or an approach for promoting long-term compliance of these interventions. The objective of this proposal is to identify the optimal approach to FMS self-management. The study is a randomized, controlled trial comparing coping skills training (the Arthritis Foundation Fibromyalgia Self-Help Course (FSHC)) with two exercise programs - cardiovascular and flexibility training with and without strength training - and a combination (the FSHC plus the strength training exercise program). Each intervention period will last 16 weeks and include group sessions led by trained personnel. Subjects will be followed for 6 months after completing the intervention to evaluate the short-term effect of each program. At 6 months, subjects will be randomized into two groups-one group will receive a 4 week refresher course of their original intervention every 6 months and the other group will receive no further intervention. Long-term follow up will be for 24 months after completing the 16 week intervention period. Subjects will include 200 women (four groups of 50), 25 to 65 years old with a confirmed diagnosis of FMS. Participants will undergo blinded assessment at the Beth Israel Deaconess Medical Center's GCRC at five time points-baseline, completion of the 16-week intervention and 6, 12 and 24 month follow up. We will assess health and functional status (FIQ, SF36), symptom severity (FIQ, SF36, Beck scales), self-efficacy (Arthritis Self-Efficacy Scale), fitness (muscle strength, cardiovascular fitness, flexibility) and health care utilization (direct and indirect costs). The study will improve treatment outcomes for persons with FMS by identifying the optimal self-management program.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25 to 75 years of age
* A confirmed diagnosis of FMS by a primary care physician (and rheumatologist if present) using the American College of Rheumatology criteria
* Currently under care for their FMS by a primary care physician or rheumatologist
* Determined to be medically stable by their primary care physician and capable of participation in a supervised program of low to moderate intensity exercise
* Willingness to commit to time and travel requirements of project

Exclusion Criteria:

* Do not fulfill ACR definition of FMS
* Presence of a concurrent condition that limits a person's ability to perform the exercise program (i.e., advanced RA or OA, recent MI)
* History of a positive exercise/stress test, or current cardiovascular, pulmonary, neurological, or renal disease where an exercise program is contraindicated
* Uncontrolled hypertension, diabetes, asthma, or heart failure
* Physician does not want his/her patient to participate for any reason

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2002-10-10 (Actual); Primary Completion 2005-09-21 (Actual); Study Completion 2005-09-21 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | Baseline, 16 wks and 10 months

SECONDARY OUTCOMES:
SF36 subscales | Baseline, 16 wks and 10 months
Beck Depression Inventory | Baseline, 16 wks and 10 months
Beck Anxiety Inventory | Baseline, 16 wks and 10 months
6 minute Walk Test | Baseline, 16 wks and 10 months
1 Repetition Maximum Chest Press | Baseline, 16 wks and 10 months
1 Repetition Maximum Leg Press | Baseline, 16 wks and 10 months
Self Efficacy Scale | Baseline, 16 wks and 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Rooks, PhD, Principal Investigator — Beth Israel Deaconess Medical Center

IPD SHARING:
Plan to Share IPD: No
No plan was prepared, as no data was to be shared.

REFERENCES:
- [Background] Rooks DS, Silverman CB, Kantrowitz FG. The effects of progressive strength training and aerobic exercise on muscle strength and cardiovascular fitness in women with fibromyalgia: a pilot study. Arthritis Rheum. 2002 Feb;47(1):22-8. doi: 10.1002/art1.10180. PMID 11932874
- [Result] Rooks DS, Gautam S, Romeling M, Cross ML, Stratigakis D, Evans B, Goldenberg DL, Iversen MD, Katz JN. Group exercise, education, and combination self-management in women with fibromyalgia: a randomized trial. Arch Intern Med. 2007 Nov 12;167(20):2192-200. doi: 10.1001/archinte.167.20.2192. PMID 17998491